CLINICAL TRIAL: NCT05225337
Title: Time Restricted Eating for the Treatment of Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Krista Varady, Professor of Nutrition, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-1086
Record Dates: First submitted 2022-01-25; First posted 2022-02-04 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Diabetes Mellitus, Type 2; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Time restricted feeding (TRF) (Experimental): 8-h eating window Ad libitum food intake from 12-8 pm every day Fasting from 8-12 pm every day (16-h fast)
  Interventions: Other: Time restricted feeding (TRF)
- Daily calorie restriction (CR) (Experimental): 25% energy restriction every day Diet counseling provided
  Interventions: Other: Daily calorie restriction
- Control (No Intervention): Ad libitum food intake, eating over more than 10 hours per day

INTERVENTIONS:
Other: Time restricted feeding (TRF) — 8-h eating window Ad libitum food intake from 12-8 pm every day Fasting from 8-12 pm every day (16-h fast)
  Arms: Time restricted feeding (TRF)
Other: Daily calorie restriction — 25% energy restriction every day Diet counseling provided
  Arms: Daily calorie restriction (CR)

SUMMARY:
Innovative lifestyle strategies to treat type 2 diabetes (T2DM) are critically needed. At present, daily calorie restriction (CR) is the main diet prescribed to patients with T2DM for weight loss. However, many patients find it difficult to adhere to CR because calorie intake must be vigilantly monitored every day.

In light of these problems with CR, another approach that limits timing of food intake, instead of number of calories consumed, has been developed. This diet is called "time restricted eating" (TRE) and involves confining the period of food intake to 6-8 h per day. TRE allows individuals to self-select foods and eat ad libitum during a large part of the day, which greatly increases compliance to these protocols. Recent findings show that TRE is effective for weight loss and improved glycemic control in patients with obesity and prediabetes. However no long-term randomized controlled trial has examined whether TRE is safe and effective for patients with obesity and T2DM.

This study is a 6-month randomized, controlled trial that aims to compare the effects of TRE (eating all food between 12:00 pm to 8:00 pm, without calorie counting), versus CR (25% energy restriction daily), and a control group eating over a period of 10 or more hours per day, on change in body weight (%), glycemic control, and cardiometabolic risk factors, in adults with obesity and T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* BMI between 30 and 50 kg/m2
* Previously diagnosed with type 2 diabetes
* HbA1c between 6.5 and 11%
* Sedentary or lightly active

Exclusion Criteria:

* HbA1c below 6.5 or greater than 11%
* Have a history of cardiovascular disease
* History of eating disorders (anorexia, bulimia, or binge eating disorder)
* Not weight stable for 3 months prior to the beginning of study (weight gain or loss > 4%)
* Eating within less than a 10 hour window at baseline
* Perimenopausal (menses does not appear every 27-32d)
* Pregnant, or trying to become pregnant
* Night shift workers
* Smokers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Change in percent body weight | Measured at baseline and month 6
  Measured by an electronic scale

SECONDARY OUTCOMES:
Change in HbA1c | Measured at baseline and month 6
  Measured by outside lab (Medstar, IN)
Change in total time in euglycemic range | Measured at baseline and month 6
  Measured by continuous glucose monitor (CGM)
Change in mean glucose level | Measured at baseline and month 6
  Measured by continuous glucose monitor (CGM)
Change in standard deviation of glucose level | Measured at baseline and month 6
  Measured by continuous glucose monitor (CGM)
Change fasting glucose | Measured at baseline and month 6
  Measured by outside lab (Medstar, IN)
Change fasting insulin | Measured at baseline and month 6
  Measured by outside lab (Medstar, IN)
Change in Insulin sensitivity | Measured at baseline and month 6
  Measured as QUICKI
Change in insulin resistance | Measured at baseline and month 6
  Measured as HOMA-IR
Change in absolute body weight | Measured at baseline and month 6
  Measured by electronic scale
Change in fat mass, lean mass, visceral fat mass | Measured at baseline and month 6
  Measured by DXA
Change in waist circumference | Measured at baseline and month 6
  Measured by measuring tape
Change in body mass index (BMI) | Measured at baseline and month 6
  Calculated as kg/meter squared
Change in plasma lipids (total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides) | Measured at baseline and month 6
  Measured by outside lab (Medstar, IN)
Change in systolic and diastolic blood pressure | Measured at baseline and month 6
  Measured by blood pressure cuff
Change in heart rate | Measured at baseline and month 6
  Measured by blood pressure cuff
Change in energy and nutrient intake | Measured at baseline and month 6
  Measured by 7-day food record
Change in dietary adherence | Measured at baseline, month 3, and month 6
  Measured by 7-day food record and adherence log
Change in physical activity (steps/d) | Measured at baseline and month 6
  Measured by pedometer
Adverse events | Measured weekly from baseline to month 6
  Measured by adverse events survey
Change in medication effect score (MES) | Measured at baseline and month 6
  Measured by survey. Total score 0-100. Lower scores indicate less medication used, higher scores indicate more medication used.
Change in sleep quality | Measured at baseline and month 6
  Measured by Pittsburgh Sleep Quality Index (PSQI), total score of 0-21. A PSQI total score greater than 5 indicates poor sleep quality.
Change in insomnia severity | Measured at baseline and month 6
  Measured by Insomnia Severity Index (ISI), total score of 0-28. The total score for the ISI is interpreted as follows: no clinically significant insomnia (0-7), sub-threshold insomnia (8-14), moderate severity insomnia (15-21), and severe insomnia (22-28).
Change in risk of sleep apnea | Measured at baseline and month 6
  Measured by Berlin Questionnaire, measures proportion of participants at high risk for sleep apnea

CONTACTS AND LOCATIONS:
Overall Officials: Krista Varady, Principal Investigator — University of Illinois Chicago
Locations (1):
- University of Illinois Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pavlou V, Cienfuegos S, Lin S, Ezpeleta M, Ready K, Corapi S, Wu J, Lopez J, Gabel K, Tussing-Humphreys L, Oddo VM, Alexandria SJ, Sanchez J, Unterman T, Chow LS, Vidmar AP, Varady KA. Effect of Time-Restricted Eating on Weight Loss in Adults With Type 2 Diabetes: A Randomized Clinical Trial. JAMA Netw Open. 2023 Oct 2;6(10):e2339337. doi: 10.1001/jamanetworkopen.2023.39337. PMID 37889487